CLINICAL TRIAL: NCT03948438
Title: Clinical Outcome of Endoscopic Treatment for Zenker's Diverticulum
Brief Title: Endoscopic Treatment for Zenker's Diverticulum
Status: Recruiting | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: ICH Zenker
Record Dates: First submitted 2019-05-08; First posted 2019-05-14 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Zenker Diverticulum
MeSH Terms: conditions — Zenker Diverticulum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endoscopic septotomy — Patients will be placed in left lateral decubitus position, either in conscious sedation or under deep sedation with propofol or endotracheal intubation.The procedure will be performed with a flexible standard endoscope and started with initial endoscopic examination with suction of possible retained material insidethe diverticulum. An incision of the bridge between the ZD and the esophagus will be done (using one endoscopic procedure as POES or FESD or other)

SUMMARY:
Zenker's diverticulum (ZD) is a rare benign condition, due to an acquired sac-like outpouching of the mucosa and submucosa layers originating from the pharyngoesophageal junction. Endoscopic techniques like flexible endoscopic septum division (FESD) or per-oral endoscopic septotomy (POES), represent a minimally invasive alternative to surgery or to rigid endoscopic procedure to treat ZD. The goal of the research will be to evaluate the safety of the procedures and to measure Zenker-symptom severity in all patients treated by endoscopic procedures.

ELIGIBILITY:
Inclusion Criteria:

* patients with symptomatic ZD treated by endoscopic procedures

Exclusion Criteria:

* pregnancy and breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients affected by ZD and treated by endoscopic procedures.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2009-01-01 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | 24 hours after the procedure
  Any complications as bleeding, perforation, others

SECONDARY OUTCOMES:
symptoms after the procedure | up to 5 years
  The frequency of symptoms such as dysphagia, regurgitation, weight loss

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Research Hospital, Rozzano, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Repici A, Cappello A, Spadaccini M, Nicoletti R, Carrara S, Fugazza A, Galtieri PA, Lamonaca L, Romana C, Badalamenti M, Di Leo M, Pellegatta G, Ferrara EC, Anderloni A, Maselli R. Cap-Assisted Endoscopic Septotomy of Zenker's Diverticulum: Early and Long-Term Outcomes. Am J Gastroenterol. 2021 Sep 1;116(9):1853-1858. doi: 10.14309/ajg.0000000000001356. PMID 34236338